CLINICAL TRIAL: NCT06513208
Title: Ketorolac Effects on Post-operative Pain and Lumbar Fusion: a Double Blind Randomized Controlled Trial
Brief Title: Ketorolac Effects on Post-operative Pain and Lumbar Fusion
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Maryland St. Joseph Medical Center (Other)
Collaborators: Medical Metrics Diagnostics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HP-00109853
Record Dates: First submitted 2024-06-25; First posted 2024-07-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Lumbar Spinal Fusion
Keywords: ketorolac; toradol; lumbar spine fusion
MeSH Terms: interventions — Ketorolac Tromethamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Ketorolac arm (Active Comparator)
  Interventions: Drug: Ketorolac Tromethamine
- Placebo Arm (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ketorolac Tromethamine — IV Ketorolac 15mg every 6 hours, x 4 doses
  Arms: Ketorolac arm
Drug: Placebo — IV saline as placebo
  Arms: Placebo Arm

SUMMARY:
A double blind prospective randomized trial of IV ketorolac vs. placebo in management of patients undergoing lumbar one or two level spinal fusions.

ELIGIBILITY:
Inclusion Criteria:

* 18-85 years old (inclusive)
* Elective posterior lumbar instrumented fusion
* One or two level fusion
* Consent to participate in study and willing to adhere to study follow up
* English proficiency

Exclusion Criteria:

* < 18 or > 85 years old
* History of renal failure, dialysis, or creatinine over 1.50 mg/dl
* Active or recent smoker (active within past 6 months)
* Revision surgery
* Auto/worker compensation
* Active cancer or history of chemotherapy in past 6 months
* Active narcotic use within 3 months of surgery date
* Infection at operative levels
* Any allergies to NSAIDs or Opioids

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Ketorolac results in decreased post-op opioid use when administered in the first 48 hours (measured by calculating the total amount of MME utilized during the patient's inpatient stay and comparing the control and experimental groups). | 12 months

SECONDARY OUTCOMES:
Ketorolac use does not decrease spinal fusion rates in one or two level fusion (failure defined as by > than 2 degrees motion on standardized flexion/extension x-rays compared to pre-op imaging analyzed by SpineCAMP software at 6 and 12 months post-op). | 12 months
Ketorolac use decreases average length of hospital stay (length of stay for both the control group and the experimental group will be counted, and a statistical average for each group will be calculated and compared). | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland St. Joseph Medical Center, Towson, Maryland, United States

IPD SHARING:
Plan to Share IPD: No